CLINICAL TRIAL: NCT07063277
Title: Comparison of the Diagnostic Value of the Oxygen Reserve Index (ORI) and Spirometry Tests in Predicting Postoperative Respiratory Complications in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Comparison of Oxygen Reserve Index and Spirometry in Predicting Respiratory Complications After Coronary Artery Bypass Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Bilkent Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Muhammed Talha Daşgın, Anesthesiology and Reanimation Doctor, Principal Investigator, Ankara Bilkent Sehir Hastanesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ankara Bilkent City Hospital 2; TABED 1-25-1274 (Other: Ankara Bilkent City Hospital)
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Coronary Arterial Disease (CAD); Coronary Artery Bypass Graft (CABG); Postoperative Pulmonary Complication
Keywords: Postoperative Pulmonary Complications; Coronary Artery Bypass Grafting; Oxygen Reserve Index; Spirometry; Cardiac Surgery Risk Assessment
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preoperative Evaluation with ORI and Spirometry (Experimental): All participants in this arm will undergo preoperative evaluation using two non-invasive methods: the Oxygen Reserve Index (ORI) and spirometry. ORI will be measured via a fingertip pulse co-oximetry sensor, reflecting oxygen reserve within the PaO₂ range of 100-200 mmHg. Measurements will be taken during routine preoxygenation with room air and supplemental oxygen. Spirometry will be conducted according to standard pulmonary function testing protocols and will include FEV₁, FVC, and FEV₁/FVC ratio. The aim is to assess and compare the predictive value of ORI and spirometry for identifying postoperative respiratory complications in patients undergoing coronary artery bypass grafting (CABG). No therapeutic intervention will be applied.
  Interventions: Device: Preoperative Evaluation with ORI and Spirometry

INTERVENTIONS:
Device: Preoperative Evaluation with ORI and Spirometry — All participants in this single-arm diagnostic study will undergo preoperative evaluation involving two non-invasive respiratory assessment methods: the Oxygen Reserve Index (ORI) and spirometry. ORI will be measured using a multi-wavelength pulse co-oximetry sensor placed on the patient's fingertip. This sensor provides a continuous, real-time index (ranging from 0.00 to 1.00) that reflects the patient's oxygen reserve within a PaO₂ range of approximately 100-200 mmHg.
  Spirometry will be performed using standard pulmonary function testing protocols. Each patient will be instructed to perform forced expiratory maneuvers to obtain parameters including forced expiratory volume in one second (FEV₁), forced vital capacity (FVC), and the FEV₁/FVC ratio. These values will be recorded prior to surgery and interpreted according to internationally accepted reference ranges.

SUMMARY:
Coronary artery disease (CAD) is one of the most common cardiac conditions, primarily caused by atherosclerosis. Studies have shown that environmental factors such as lifestyle, diet, genetics, and air pollution contribute to the increasing prevalence of atherosclerosis. Despite advances in non-invasive and medical therapies, coronary artery bypass grafting (CABG) remains a definitive treatment in many cases. CABG is commonly performed using cardiopulmonary bypass (CPB), which increases the risk of additional complications. Among postoperative complications, pulmonary events are the most frequent and are closely associated with increased morbidity and mortality.

Postoperative pulmonary complications (PPCs) significantly raise healthcare costs, prolong hospital stays, and worsen patient outcomes. Cardiac surgery increases susceptibility to PPCs through factors such as sternotomy, CPB, myocardial protection via hypothermia, and phrenic nerve injury. These factors impair thoracic compliance, diaphragm movement, and mucociliary function. Mechanical ventilation further contributes through inflammatory responses that may cause barotrauma and volutrauma.

The incidence of PPCs varies from 1.96% to 43.7%, depending on patient characteristics, surgical type, and diagnostic criteria. With an aging population and more high-risk patients undergoing surgery, the incidence of PPCs is expected to rise. Reported preoperative risk factors include advanced age, active or recent smoking, BMI >25, heart failure, prior myocardial infarction, chronic lung disease, type 2 diabetes mellitus, hypertension, and ASA score >2. Intraoperative factors include prolonged anesthesia, CPB duration >95 minutes, multiple grafts, and use of the internal mammary artery. Postoperative contributors include prolonged ventilation, nasogastric tube use, and insufficient nursing care.

Common PPCs include atelectasis, pneumonia, bronchospasm, pulmonary embolism, pleural effusion, acute respiratory distress syndrome (ARDS), pneumothorax, hemothorax, and transfusion-related acute lung injury (TRALI). Atelectasis is observed in 30-72% of cases on postoperative chest X-rays. TRALI is the leading cause of transfusion-related death and is characterized by hypoxia and bilateral pulmonary infiltrates. Pleural effusions are associated with low BMI, female sex, atrial fibrillation, heart failure, valve surgery, and anticoagulant use. Phrenic nerve injury, often resulting from internal thoracic artery dissection or cold-induced damage during myocardial protection, leads to unilateral diaphragmatic dysfunction.

Hospital-acquired infections, particularly pneumonia, are among the most common and costly non-cardiac complications following cardiac surgery. Pneumonia occurs in 2.4%-20% of cases, while ventilator-associated pneumonia affects 35.2% of patients intubated longer than 48 hours. ARDS is the most severe PPC, involving widespread alveolar injury, endothelial disruption, and non-cardiogenic pulmonary edema. Tension pneumothorax may also occur after chest tube removal.

Spirometry is a standard preoperative test used to assess lung function, primarily through FEV₁ and FVC values. These measurements help detect obstructive or restrictive defects. FEV₁/FVC <70% has been identified as an independent risk factor for PPCs. However, spirometry's predictive value is limited. A systematic review by Dankert et al. reported sensitivities ranging from 38% to 84% and specificities from 55% to 99%. Combined data yielded a sensitivity of 62%, specificity of 70%, and an area under the curve (AUC) of 0.74.

Pulse oximetry alone cannot reliably indicate PaO₂ above 100 mmHg or provide information on oxygen reserve. The Oxygen Reserve Index (ORI) is a novel, continuous, and non-invasive parameter that evaluates oxygenation status in the mild hyperoxic range (PaO₂ 100-200 mmHg). ORI values range from 0.00 to 1.00 and correlate with changes in PaO₂. ORI >0.24 corresponds to PaO₂ ≥100 mmHg when SpO₂ exceeds 98%, while ORI >0.55 may indicate PaO₂ ≥150 mmHg. A declining ORI trend approaching 0.24, despite SpO₂ >98%, can signal impending hypoxemia.

Given the substantial impact of PPCs on postoperative outcomes and the limitations of spirometry in accurately predicting these complications, there is a need for more reliable preoperative assessment tools. The present study aims to compare the diagnostic performance of the Oxygen Reserve Index and spirometry in predicting postoperative respiratory complications in patients undergoing coronary artery bypass surgery. The goal is to identify a more accurate and effective method for preoperative pulmonary risk stratification.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is one of the most prevalent cardiac disorders caused by atherosclerosis. Comprehensive studies have shown that changes in environmental factors such as lifestyle, diet, genetics, and air pollution contribute to an increased incidence of atherosclerosis. Despite the continuous development of non-invasive and medical treatments, coronary artery bypass grafting (CABG) remains the final treatment option for many patients. In this procedure, open-heart surgery is performed with or without the use of cardiopulmonary bypass (CPB), during which vascular grafts are created. In most cases, CPB is utilized, which may lead to additional complications beyond those associated with the surgery itself. Following CABG, cardiovascular, pulmonary, renal, infectious, and psychiatric complications may occur. Among these, pulmonary complications are the most commonly encountered and are significantly associated with morbidity and mortality.

Postoperative pulmonary complications (PPCs) following cardiac surgery increase healthcare costs, prolong hospital stay, and elevate morbidity and mortality rates. Cardiac surgery predisposes to PPCs more than other surgical types due to median sternotomy/thoracotomy, CPB, myocardial protection via hypothermia, and phrenic nerve injury. It directly impairs thoracic compliance, diaphragm function, and mucociliary clearance. Additionally, mechanical ventilation activates local and systemic inflammatory responses, leading to volutrauma and barotrauma.

The incidence of PPCs following cardiac surgery ranges from 1.96% to 43.7%, depending on patient-related risk factors, the type of cardiac procedure performed, and the definition of PPC used. With the increasing number of high-risk patients undergoing cardiac surgery due to an aging population, a rise in PPC incidence is expected. Preoperative risk factors identified in various studies include age above 65 or 80 years, active smoking within the past 6 or 12 months, body mass index over 25, heart failure, history of myocardial infarction (MI), chronic lung disease, type 2 diabetes mellitus (DM2), hypertension (HT), and an American Society of Anesthesiologists (ASA) score greater than 2. Intraoperative risk factors include anesthesia duration longer than 270 minutes, CPB duration longer than 95 minutes, repair of four or more vessels, and use of the internal mammary artery (IMA) as a graft. Postoperative risk factors include mechanical ventilation for more than 10 hours, presence of a nasogastric tube, and lack of high-quality nursing care.

PPCs include atelectasis, pneumonia, bronchospasm, pulmonary embolism, pleural effusion, acute respiratory distress syndrome (ARDS), pneumothorax, hemothorax, mechanical ventilation longer than 48 hours, transfusion-related acute lung injury (TRALI), and phrenic nerve injury. Atelectasis is a common cause of hypoxemia and impaired gas exchange following cardiac surgery. Postoperative chest X-rays show atelectasis in 30-72% of patients, making it one of the leading causes of respiratory dysfunction. TRALI is the most common transfusion-related adverse event and the leading cause of transfusion-related deaths globally. It is characterized by acute hypoxia and bilateral pulmonary infiltrates following allogeneic blood transfusion. Pleural effusions after CABG are associated with low body mass index, female sex, history of atrial fibrillation, heart failure, concomitant valve surgery, and anticoagulant use. Surgical injury to the phrenic nerve often results in unilateral loss of diaphragmatic function and is commonly observed during dissection of the internal thoracic artery. Previous studies have shown that phrenic nerve injury may also occur due to cold exposure during myocardial protection strategies.

Healthcare-associated infections are a leading cause of non-cardiac morbidity after cardiac surgery. Among these, pneumonia is the most frequently observed, the most expensive, and the most resource-intensive infection. Pneumonia develops in 2.4% to 20% of patients following cardiac surgery. Additionally, ventilator-associated pneumonia occurs in 35.2% of patients who remain on mechanical ventilation for more than 48 hours. ARDS is the most severe pulmonary complication after cardiac surgery, characterized by pro-inflammatory injury to the alveolar structure, widespread endothelial damage, severe hypoxia, and non-cardiogenic pulmonary edema.

Mediastinal and pleural drains are commonly placed after cardiac surgery and are removed when fluid output is minimal and hemodynamic stability is achieved. However, recurrence due to tension pneumothorax following drain removal represents a life-threatening complication. This occurs when a one-way air flow between the lung parenchyma and the pleural space causes air to become trapped in the pleural cavity.

Spirometry is used to assess pulmonary function and is a widely accepted preoperative test in thoracic surgeries. It evaluates the forced expiratory volume in one second (FEV₁) and forced vital capacity (FVC), aiding in the diagnosis of obstructive or restrictive ventilatory defects. Spirometry is closely associated with chronic obstructive pulmonary disease (COPD), asthma, and interstitial lung diseases. An FEV₁/FVC ratio below 70% is considered an independent risk factor for postoperative complications in thoracic surgeries.

Although spirometry is a conventional respiratory function test, its sensitivity and specificity in predicting PPCs remain suboptimal. A systematic review by Dankert et al. reported sensitivities ranging from 38% to 84% and specificities from 55% to 99%. Based on the pooled data from the included studies, a ROC analysis was performed to assess spirometry's predictive value for PPCs. The average sensitivity was found to be 62%, specificity 70%, and area under the curve (AUC) 0.74.

While pulse oximetry is a standard monitoring tool, it does not reliably indicate whether PaO₂ exceeds 100 mmHg or whether oxygen reserves are increasing. Therefore, the Oxygen Reserve Index (ORI) may assist in identifying inadequate preoxygenation and provide preliminary information on pulmonary oxygen reserve. ORI is a non-invasive and continuous parameter that evaluates real-time oxygen reserve within a mild hyperoxic range (approximately PaO₂ 100-200 mmHg). It is measured using a finger sensor and varies between 0.00 and 1.00 depending on oxygen reserve status. Changes in ORI values reflect corresponding changes in PaO₂ within this range. Although ORI and PaO₂ do not show exact correspondence, a positive correlation has been observed within the specified range. Studies have shown that when SpO₂ exceeds 98%, an ORI >0.24 may indicate PaO₂ ≥100 mmHg. Similarly, an ORI >0.55 appears to correspond with PaO₂ ≥150 mmHg. A decline in ORI toward 0.24 while SpO₂ remains >98% may serve as an early indicator of PaO₂ approaching 100 mmHg.

Given the high morbidity and mortality associated with PPCs, especially in cardiac surgery cases, accurate preoperative prediction and appropriate risk stratification are of critical importance. Due to the limited predictive power of spirometry alone, there is a need for novel and updated approaches. The current study aims to evaluate the effectiveness of ORI and spirometry in predicting PPCs. Based on the findings, a more effective method for anticipating pulmonary complications in cardiac surgery may be developed.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective coronary artery bypass grafting (CABG) surgery.
* Aged 18 years or older at the time of enrollment.
* Provided written informed consent to participate in the study.
* Medically stable and cooperative for preoperative respiratory assessments (ORI and spirometry).

Exclusion Criteria:

* Refusal to participate or failure to provide informed consent.
* Age under 18 years.
* Left ventricular ejection fraction below 40% on preoperative evaluation.
* Presence of cognitive impairment or psychiatric disorders preventing cooperation (e.g., dementia, Alzheimer's disease).
* Severe anemia defined as hemoglobin level below 8 g/dL.
* Undergoing emergency surgery rather than elective CABG.
* Anatomical or mechanical obstruction that may impair nasal oxygenation (e.g., severe nasal septum deviation, presence of a nasogastric tube).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Respiratory Complications | Postoperative 48 hours
  Postoperative respiratory complications, including but not limited to collapse of part or all of a lung (atelectasis), lung infection (pneumonia), the need for continued use of a breathing machine for an extended period after surgery (prolonged mechanical ventilation), or abnormalities in oxygen levels in the blood (oxygenation disorders), will be systematically assessed during the first 48 hours following the surgical procedure. Each event will be evaluated based on clinical symptoms such as shortness of breath, abnormal breath sounds, or decreased oxygen saturation. Additional confirmation will be obtained through diagnostic tools including chest imaging (such as chest X-ray), arterial blood gas analysis, and ventilator parameters. The presence, timing, and severity of each complication will be documented, as well as any medical or mechanical respiratory support required (such as supplemental oxygen, non-invasive ventilation, or reintubation)

SECONDARY OUTCOMES:
Preoperative Peak ORI Value | Preoperative period (within 24 hours prior to surgery)
  The highest Oxygen Reserve Index (ORI) value recorded during the preoxygenation phase will be measured using a multi-wavelength fingertip pulse co-oximetry sensor. The ORI value (ranging from 0.00 to 1.00) reflects the patient's oxygen reserve within a PaO₂ range of approximately 100-200 mmHg. This parameter will be used to investigate the association between preoperative oxygen reserve and the risk of postoperative respiratory complications.
FEV₁ (Forced Expiratory Volume in 1 second) | Preoperative period (within 24 hours prior to surgery)
  The volume of air forcefully exhaled during the first second of a forced breath, measured preoperatively via standardized spirometry. FEV₁ serves as a primary indicator of airway obstruction and overall pulmonary function. Both absolute values and corresponding z-scores (adjusted for age, sex, height, and ethnicity) will be recorded to enable individualized interpretation and comparison. These values will be used to evaluate baseline pulmonary status and its association with postoperative respiratory complications.
Intraoperative Respiratory Complications | During surgery
  Respiratory complications occurring intraoperatively will be documented in real-time by the anesthesia team. These may include bronchospasm, desaturation events (SpO₂ < 90%), unexpected need for endotracheal intubation, or intraoperative airway management difficulties. Each event will be classified according to timing, severity, and the intervention required.
Intraoperative Hemodynamic or Surgical Complications | During surgery
  This outcome includes any intraoperative complications unrelated to the respiratory system, such as low blood pressure requiring the use of medications to support circulation (mean arterial pressure below 65 millimeters of mercury), abnormal heart rhythms, bleeding that requires transfusion of blood or blood products, technical difficulties during the connection of bypass grafts, or prolonged duration of the heart-lung machine use. All events will be categorized based on their type and severity.
Duration of Intensive Care Unit and Total Hospital Stay | From the date of surgery until ICU and hospital discharge, assessed up to 180 days
  The total number of full calendar days each participant remains in the intensive care unit after surgery, as well as the total length of hospitalization from the date of surgery until discharge from the hospital, will be recorded. These durations will serve as indicators of early and overall postoperative recovery. The results will be analyzed in relation to preoperative respiratory assessments, including Oxygen Reserve Index and spirometry measurements. This outcome will also provide insight into healthcare resource utilization and patient stratification based on preoperative respiratory function.
In-Hospital Postoperative Mortality | From the date of surgery until hospital discharge, assessed up to 180 days
  Any death occurring during the same hospital admission after the surgical procedure will be recorded and classified based on time of occurrence and primary cause. This outcome will be used to assess the relationship between baseline respiratory parameters and mortality risk.
FVC (Forced Vital Capacity) | Preoperative period (within 24 hours prior to surgery)
  The total volume of air exhaled forcefully after a maximal inhalation, assessed through preoperative spirometry. FVC reflects pulmonary capacity and is essential in identifying restrictive ventilatory defects. Both raw FVC values and corresponding z-scores will be recorded. This parameter will contribute to assessing baseline lung mechanics and stratifying risk for postoperative respiratory dysfunction.
PEF (Peak Expiratory Flow) | Preoperative period (within 24 hours prior to surgery)
  The maximum flow rate achieved during the forced expiratory maneuver, representing large airway patency and expiratory effort. PEF will be measured preoperatively using spirometry, with both raw values and z-scores recorded. It provides insight into expiratory muscle function and airway resistance, potentially correlating with postoperative respiratory recovery and complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scheeren TWL, Belda FJ, Perel A. The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):379-389. doi: 10.1007/s10877-017-0049-4. Epub 2017 Aug 8. PMID 28791567
- [Result] Chen ST, Min S. Oxygen reserve index, a new method of monitoring oxygenation status: what do we need to know? Chin Med J (Engl). 2020 Jan 20;133(2):229-234. doi: 10.1097/CM9.0000000000000625. PMID 31904726
- [Result] Dankert A, Dohrmann T, Loser B, Zapf A, Zollner C, Petzoldt M. Pulmonary Function Tests for the Prediction of Postoperative Pulmonary Complications. Dtsch Arztebl Int. 2022 Feb 18;119(7):99-106. doi: 10.3238/arztebl.m2022.0074. PMID 34939921
- [Result] Yoshimi K, Oh S, Suzuki K, Kodama Y, Sekiya M, Seyama K, Fukuchi Y. Impact of Airflow Limitation on Comorbidities and Postoperative Complications in Patients Undergoing Thoracic Surgery: A Retrospective Observational Study. Ann Thorac Cardiovasc Surg. 2016 Jun 20;22(3):146-52. doi: 10.5761/atcs.oa.15-00301. Epub 2016 Mar 1. PMID 26935262
- [Result] Park HJ, Kim SM, Kim HR, Ji W, Choi CM. The value of preoperative spirometry testing for predicting postoperative risk in upper abdominal and thoracic surgery assessed using big-data analysis. J Thorac Dis. 2020 Aug;12(8):4157-4167. doi: 10.21037/jtd-19-2687. PMID 32944327
- [Result] Tanner TG, Colvin MO. Pulmonary Complications of Cardiac Surgery. Lung. 2020 Dec;198(6):889-896. doi: 10.1007/s00408-020-00405-7. Epub 2020 Nov 11. PMID 33175990
- [Result] Jensen L, Yang L. Risk factors for postoperative pulmonary complications in coronary artery bypass graft surgery patients. Eur J Cardiovasc Nurs. 2007 Sep;6(3):241-6. doi: 10.1016/J.EJCNURSE.2006.11.001. Epub 2007 Mar 7. PMID 17347049
- [Result] Thanavaro J, Taylor J, Vitt L, Guignon MS, Thanavaro S. Predictors and outcomes of postoperative respiratory failure after cardiac surgery. J Eval Clin Pract. 2020 Oct;26(5):1490-1497. doi: 10.1111/jep.13334. Epub 2019 Dec 25. PMID 31876045
- [Result] Mali S, Haghaninejad H. Pulmonary complications following cardiac surgery. Arch Med Sci Atheroscler Dis. 2019 Dec 31;4:e280-e285. doi: 10.5114/amsad.2019.91432. eCollection 2019. PMID 32368683